CLINICAL TRIAL: NCT00790244
Title: A Scandinavian Sarcoma Group Treatment Protocol for Adult Patients With Non-metastatic High-risk Soft Tissue Sarcoma of the Extremities and Trunk Wall
Brief Title: A Scandinavian Sarcoma Group Protocol for Patients With High-risk Soft Tissue Sarcoma of the Extremities and Trunk Wall
Acronym: SSGXX
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Oslo University Hospital (Other)
Collaborators: Scandinavian Sarcoma Group (Other)
Responsible Party: Kirsten Sundby Hall, Rikshospitalet-Radiumhospitalet HF
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT number 2007-001152-39
Record Dates: First submitted 2008-11-12; First posted 2008-11-13 (Estimated); Last update posted 2011-07-06 (Estimated); Status verified 2008-11

CONDITIONS: Soft Tissue Sarcoma; Non Metastatic Disease
Keywords: Soft-tissue sarcomas; prognostic factors; adjuvant; chemotherapy; radiotherapy; metastases-free survival; toxicity; High malignancy grade; High-risk for metastases; Adult
MeSH Terms: conditions — Sarcoma | interventions — Doxorubicin; Ifosfamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm 2 (Experimental): <70y: 6 cycles with doxorubicin 60mg/m2+ifosfamide 6g/m2 of each 21day cycle and radiotherapy 36Gy (1.8Gy per fraction, two fractions daily) will be given between cycle 3 and 4.
  (>=70y: doxorubicin 50mg/m2+ifosfamide 5g/m2)
  Interventions: Drug: doxorubicin , ifosfamide; Drug: doxorubicin, ifosfamide
- Arm 3 (Experimental): <70y: 6 cycles with doxorubicin 60mg/m2+ifosfamide 6g/m2 of each 21day cycle and radiotherapy 45Gy (1.8Gy per fraction, two fractions daily) will be given between cycle 3 and 4.
  (>=70y: doxorubicin 50mg/m2+ifosfamide 5g/m2)
  Interventions: Drug: doxorubicin , ifosfamide
- Group B (Experimental): <70y: 6 cycles with doxorubicin 60mg/m2+ifosfamide 6g/m2 of each 21day cycle and radiotherapy 36Gy (1.8Gy per fraction, two fractions daily) will be given between cycle 2 and 3.
  (>=70y: doxorubicin 50mg/m2+ifosfamide 5g/m2)
  Interventions: Drug: doxorubicin , ifosfamide; Drug: doxorubicin, ifosfamide
- Arm 1 (Experimental): <70y: 6 cycles with doxorubicin 60mg/m2+ifosfamide 6g/m2 of each 21day cycle (>=70y: doxorubicin 50mg/m2+ifosfamide 5g/m2)
  Interventions: Drug: doxorubicin , ifosfamide; Drug: doxorubicin, ifosfamide

INTERVENTIONS:
Drug: doxorubicin , ifosfamide — doxorubicin 60mg/m2+ifosfamide 6g/m2 every third week
  Other Names: Doxorubicin; Holoxan
Drug: doxorubicin, ifosfamide — Doxorubicin and Ifosfamide given every three weeks, totally 6 courses.
  Other Names: Doxorubicin; Holoxan
  Arms: Arm 1
Drug: doxorubicin, ifosfamide — <70y: 6 cycles with doxorubicin 60mg/m2+ifosfamide 6g/m2 of each 21day cycle and radiotherapy 36Gy (1.8Gy per fraction, two fractions daily) will be given between cycle 3 and four.
  (>=70y: doxorubicin 50mg/m2+ifosfamide 5g/m2)
  Other Names: Doxorubicin; Holoxan
  Arms: Arm 2
Drug: doxorubicin, ifosfamide — <70y: 6 cycles with doxorubicin 60mg/m2+ifosfamide 6g/m2 of each 21day cycle and radiotherapy 36Gy (1.8Gy per fraction, two fractions daily) will be given between cycle 2 and 3.
  (>=70y: doxorubicin 50mg/m2+ifosfamide 5g/m2)
  Other Names: Doxorubicin; Holoxan
  Arms: Group B

SUMMARY:
SSG XX is a phase II trial for high-risk soft tissue sarcomas (STS) of the extremities and trunk wall. Prognostic factors (histopathological markers) are used to identify high-risk tumors. SSG XX will evaluate chemo- and radiotherapy given adjuvantly to these patients. In a specified group of patients also preoperatively given therapy will be studied.

DETAILED DESCRIPTION:
SSG XX, the third adjuvant STS protocol by SSG, is a phase II non-randomized trial in patients with high risk to develop metastases. SSG XX is based on a previous SSG trial (SSG XIII) regarding use of prognostic markers to identify high-risk tumors and include very similar chemo- and radiotherapy treatment schedules compared to SSG XIII, but the new protocol also includes a treatment arm with preoperative chemo- and radiotherapy for patients with an obvious risk for intralesional surgery initially.

Patients: In this new adjuvant protocol SSG adopts an inclusion decision algorithm based on the following criteria: 1.vascular invasion or 2. presence of at least two of the risk factors: tumor size =>8 cm, necrosis or infiltrative growth(all defined microscopically by the pathologist. The system was developed retrospectively by evaluation of 434 primary histologically high grade (III-IV) STS from the SSG registry, and was later validated in a series of 175 patients in which patients with a high risk for metastases (>40 %) and low risk (<15 %) were separated (Engellau J et al.Eur J Ca 2007 43: 1927-34). Inclusion criteria: age ≥ 18 y and <75 y. Primary end point is metastasis-free survival. Local recurrence and toxicity will also be studied.

Treatment: Six cycles of doxorubicin 60mg/m2 and ifosfamide 6g/m2 will be given adjuvantly (to patients ≥ 70y: 50mg/m2 and 5g/m2 ). Dependent on surgical resection margins, 36Gy or 45Gy (1,8Gy per fraction, two fractions daily) will be given interpolated with chemotherapy.

Conclusion: SSG XX will evaluate chemo-and radiotherapy given adjuvantly to patients with STS and high risk for metastases (arm A). In a specified group of patients also preoperatively given therapy will be studied(arm B). Other sarcoma centers are invited to participate in the study.

ELIGIBILITY:
Inclusion Criteria:

Group A: Histological high-grade malignancy soft tissue sarcomas of the extremity and trunk wall.

Patients fulfilling the high-risk criteria defined above (see detailed description) Group B: Patients with histological high-grade malignancy soft tissue sarcomas of the extremity and trunk wall for whom surgery carries an obvious risk of intralesional margin

Other inclusion criteria for therapy group A and group B

* Age ≥ 18 y and ≤ 75 y
* WHO grade 0-1
* Adequate cardiac function (LVEF ≥ 50%)
* Normal GFR (clearance)
* Adequate haematologic and liver function
* All histotypes except those listed below

Exclusion Criteria:

The following histological types:

* Extraskeletal osteosarcoma and - chondrosarcoma, Ewing/PNET, rhabdomyosarcoma, Kaposi´s sarcoma, malignant mesenchymoma, clear cell sarcoma, alveolar soft part sarcoma, epithelioid sarcoma
* Radiation induced sarcoma
* No previous anthracycline treatment
* Less than 5 years free of another primary malignancy
* More than 12 weeks have elapsed since primary surgery (Group A)
* More than 4 weeks from diagnostic biopsy to start of chemotherapy (Group B)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 188 (Estimated)
Dates: Start 2007-10; Primary Completion 2012-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Metastases-free survival | time frame from start of treatment until the events metastases or death of any cause

SECONDARY OUTCOMES:
cumulative incidence of local recurrence,overall survival,acute and late toxicity,secondary malignancies | for ten years from start of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten Sundby Hall, MD,PhD, Principal Investigator — c/o: Scandinavian Sarcoma Group, Southern Swedish Regional Tumor Registry, Lund University Hospital, SE-221 85 Lund
Locations (2):
- Sweden (2):
  - Scandinavian Sarcoma Group centers, Lund, Lund
  - Scandinavian Sarcoma Group Secretariat, Lund University Hospital, Lund

REFERENCES:
- [Background] Engellau J, Samuelsson V, Anderson H, Bjerkehagen B, Rissler P, Sundby-Hall K, Rydholm A. Identification of low-risk tumours in histological high-grade soft tissue sarcomas. Eur J Cancer. 2007 Sep;43(13):1927-34. doi: 10.1016/j.ejca.2007.05.018. Epub 2007 Jul 12. PMID 17627813
- [Background] Engellau J, Bendahl PO, Persson A, Domanski HA, Akerman M, Gustafson P, Alvegard TA, Nilbert M, Rydholm A. Improved prognostication in soft tissue sarcoma: independent information from vascular invasion, necrosis, growth pattern, and immunostaining using whole-tumor sections and tissue microarrays. Hum Pathol. 2005 Sep;36(9):994-1002. doi: 10.1016/j.humpath.2005.07.008. PMID 16153463
- [Derived] Hall KS, Bruland OS, Bjerkehagen B, Lidbrink E, Jebsen N, Hagberg H, Papworth K, Hagberg O, Trovik C, Bauer H, Eriksson M. Preoperative accelerated radiotherapy combined with chemotherapy in a defined cohort of patients with high risk soft tissue sarcoma: a Scandinavian Sarcoma Group study. Clin Sarcoma Res. 2020 Nov 17;10(1):22. doi: 10.1186/s13569-020-00145-5. PMID 33292545
- [Derived] Sundby Hall K, Bruland OS, Bjerkehagen B, Zaikova O, Engellau J, Hagberg O, Hansson L, Hagberg H, Ahlstrom M, Knobel H, Papworth K, Zemmler M, Goplen D, Bauer HCF, Eriksson M. Adjuvant chemotherapy and postoperative radiotherapy in high-risk soft tissue sarcoma patients defined by biological risk factors-A Scandinavian Sarcoma Group study (SSG XX). Eur J Cancer. 2018 Aug;99:78-85. doi: 10.1016/j.ejca.2018.05.011. Epub 2018 Jun 19. PMID 29929092
- See also: Scandinavian Sarcoma Group — http://www.ssg-org.net